CLINICAL TRIAL: NCT02267460
Title: A Phase 3b, Open-label Pilot Study to Evaluate the Safety and Effectiveness of up to Four Treatment Cycles of AA4500 in Combination With the ErecAid® Esteem® Manual Vacuum Therapy System in Men With Peyronie's Disease
Brief Title: An Open-label Study to Assess the Safety and Effectiveness of AA4500 in Combination With the ErecAid® Esteem® Manual Vacuum Therapy System in Treating Men With Peyronie's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-807
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's disease; penile plaque; penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 with investigator modeling and vacuum therapy (Active Comparator): AA4500 with investigator modeling and home use of the ErecAid® Esteem® Manual Vacuum Therapy System.
  Interventions: Biological: AA4500; Device: ErecAid® Esteem® Manual Vacuum Therapy System; Procedure: Investigator Modeling
- AA4500 without investigator modeling/with vacuum therapy (Active Comparator): AA4500 without investigator modeling but with home use of the ErecAid® Esteem® Manual Vacuum Therapy System.
  Interventions: Biological: AA4500; Device: ErecAid® Esteem® Manual Vacuum Therapy System

INTERVENTIONS:
Biological: AA4500
  Other Names: Xiaflex; Xiapex; collagenase clostridium histolyticum
Device: ErecAid® Esteem® Manual Vacuum Therapy System
Procedure: Investigator Modeling
  Arms: AA4500 with investigator modeling and vacuum therapy

SUMMARY:
Enrollment will include approximately 30 AA4500 naïve subjects. Subjects will be divided by degree of penile curvature and then randomized in a 1:1 ratio to one of the following treatment groups:

* AA4500 with investigator modeling
* AA4500 without investigator modeling

Each subject will receive 2 injections of AA4500, separated by approximately 24 hours to 72 hours, repeated after 42 days (± 5 days) for up to 4 treatment cycles.

Approximately 14 days after the second injection of AA4500, each subject will visit the study site and the investigator will assess the subject and instruct the subject on appropriate use of the ErecAid® Esteem® Manual Vacuum Therapy System.

ELIGIBILITY:
Inclusion Criteria:

* Be a male ≥ 18 years of age
* Have symptom(s) of Peyronie's disease and have evidence of stable disease as determined by the investigator
* Have penile curvature of at least 30° in the dorsal, lateral, or dorsal/lateral plane at screening. It must be possible to delineate the single plane of maximal curvature for evaluation during the study
* Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile
* Voluntarily sign and date an informed consent agreement approved by the Independent Ethics Committee (IEC).
* Be able to read, complete and understand the various rating instruments in English.

Exclusion Criteria:

* Has a penile curvature of less than 30° or greater than 90° at the screening visit
* Has any of the following conditions:

  * Chordee in the presence or absence of hypospadias
  * Thrombosis of the dorsal penile artery and/or vein
  * Infiltration by a benign or malignant mass resulting in penile curvature
  * Infiltration by an infectious agent, such as lymphogranuloma venereum
  * Ventral curvature from any cause
  * Presence of an active sexually transmitted disease
  * Known active hepatitis B or C
  * Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
* Has a history of spontaneous priapism (ie, erection that lasts more than four hours)
* Has previously undergone surgery for Peyronie's disease
* Fails to have an erection which, in the opinion of the investigator, is sufficient to accurately measure the subject's penile deformity after administration of prostaglandin E1
* Has a calcified plaque as evident by appropriate radiographic evaluation, penile ultrasound that would prevent proper injection of study medication. Non-contiguous stippling of calcium is acceptable for inclusion provided the calcium deposit does not interfere with the injection of AA4500 into the plaque
* Has an isolated hourglass deformity of the penis
* Has the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of the local anesthetic would interfere with the injection of AA4500 into the plaque
* Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
* Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [>500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti-inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
* Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6-month period before screening or plans to have ESWT at any time during the study
* Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices (except for that prescribed by protocol) at any time during the study
* Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices (except for that prescribed by protocol) at any time during the study
* Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
* Has a penile Duplex Doppler ultrasound evaluation at screening that shows compromised penile hemodynamics that in the opinion of the investigator is clinically significant
* Has uncontrolled hypertension, as determined by the investigator
* Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
* Has sickle cell trait or disease, multiple myeloma, Hodgkin's lymphoma, and/or a blood dyscrasia that carries the risk for clotting or priapism
* Has an impairment of the hand(s) that would prevent safe use of the vacuum pump, as determined by the investigator
* Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
* Has received an investigational drug or treatment within 30 days before the first dose of study drug
* Has a known allergy to collagenase or any other excipient of AA4500
* Has a known allergy to any concomitant medication required as per the protocol
* Has a coagulation disorder
* Is taking a medication for chronic anticoagulation (except for ≤ 150 mg aspirin daily)
* Has received any collagenase treatments within 30 days of the first dose of study drug
* Has, at any time, received AA4500 for the treatment of Peyronie's disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percent in improvement from baseline in penile curvature | 36 Weeks
  measurement of erect penis at day 42 (cycle 2), day 84 (cycle 3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)

SECONDARY OUTCOMES:
Change in Peyronies disease bother | 36 Weeks
  Questionnaire at Day 168 (follow up 1) and day 252 (follow up 2)
Change in Peyronies disease physical symptoms | Week 36
  measurement of erect penis at day 42 (cycle 2), day 84 (cycle 3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)
Change in Peyronies disease psychological symptoms | 36 Weeks
  Questionnaire at Day 168 (follow up 1) and day 252 (follow up 2)
Change in penile plaque consistency | 36 Weeks
  Flaccid penile exam at day 42 (cycle 2), day 84 (cycle 3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)
Change in penile length | 36 Weeks
  Flaccid penile exam at day 42 (cycle 2), day 84 (cycle 3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)
Change in Peyronies disease penile pain | 36 Weeks
  examination for pain done on day 42 (cycle 2), day 84 (cycle 3), day 126 (cycle 4), day 168 (follow up visit 1) and day 252 (follow up visit 2)
A responder analysis based on subject global assessment | 36 Weeks
  Questionnaire at Day 168 (follow up 1) and day 252 (follow up 2)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Shusterman, MD, Study Director — Endo
Locations (1):
- Hospital of St John and St Elizabeth, London, United Kingdom

REFERENCES:
- [Derived] Ralph DJ, Abdel Raheem A, Liu G. Treatment of Peyronie's Disease With Collagenase Clostridium histolyticum and Vacuum Therapy: A Randomized, Open-Label Pilot Study. J Sex Med. 2017 Nov;14(11):1430-1437. doi: 10.1016/j.jsxm.2017.08.015. Epub 2017 Sep 30. PMID 28974406